CLINICAL TRIAL: NCT06789315
Title: Randomized Controlled Trial of Mycophenolate Mofetil Versus Steroid Therapy in Alcoholic Hepatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Alcoholic Hepatitis-04
Record Dates: First submitted 2025-01-13; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Mycophenolic Acid; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mycophenolate mofetil (Experimental): Intervention arm in the study will receive MMF at a dose of 750 mg twice daily for a period of 28 days.
  Interventions: Drug: Mycophenolate Mofetil
- Steroid prednisolone (Active Comparator): steroid at a dose of 40 mg for 28 days.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Mycophenolate Mofetil — MMF at a dose of 750 mg twice daily for a period of 28 days,
  Arms: mycophenolate mofetil
Drug: Prednisone — Prednisone at a dose of 40 mg for 28 days.
  Arms: Steroid prednisolone

SUMMARY:
Patients with acute alcoholic hepatitis will be identified based on national institute on alcohol abuse and alcoholism (NIAAA) will be identified, MELD score will be calculated, patents with MELD score between 20-35 will be randomized to two groups. Group A (intervention arm) will be receiving Mycofenolate mofetil at a dose of 750 mg twice daily and group B will be receiving steroid as per existing guidelines in a dose of 40 mg per day. Both the groups will be followed up for 90 days with assessment done at 4th, 7th and 28th day. Any significant event in addition will also be noted. Patients in group A will be also be monitored for development of complications like cytopenia due to Mycofenolate mofetil and infections will be monitored in both groups. Steroids will be stopped in the non-responders in group B based on Lille score at 4th and 7th day. The outcome variables of interest and to be measured are survival at 28 days and 90 days, clinical outcomes, including hospitalization and liver related outcomes.

DETAILED DESCRIPTION:
Study Design: Single-center, randomized control trial of 1 year duration.

Aim and Objective - To compare the efficacy and safety of Mycophenolate Mofetil (MMF) versus steroid therapy for the treatment of alcoholic hepatitis.

Hypothesis -

- MMF as a first line agent maybe associated with better 28 day and 90-day survival without increasing the risk of infection.

Study population: Patients > 18 years of age.Who are diagnosed as Alcoholic hepatitis based on NIAAA criteria.

* Study design: Randomized double blinded study.
* Study period: 1 year.
* Intervention: Intervention arm in the study will receive MMF at a dose of 750 mg twice daily for a period of 28 days, while the control arm will receive steroid at a dose of 40 mg for 28 days. However, based on Lille's score the decision to continue or discontinue steroid will be taken. In case of discontinuation of the drug in either group, they will be provided best medical care and nutrition as salvage therapy.
* Monitoring and assessment: History of all patients with special emphasis to alcoholic history will be taken. The diagnosis of alcoholic hepatitis is confirmed by NIAAA criteria. Liver biopsy will be done in clinically indicated cases. Patients will be classified into acute on chronic liver disease (ACLF) based on APASL criteria. Patients who are eligible for steroid therapy will be randomized to receive steroid or MMF based on computer software. Patients who are in MMF group will receive 750 mg twice daily of MMF. Patients who are in steroid group will receive 40 mg Prednisolone. The study is open label randomized control trial. Lilles score is calculated at 5th day to see for response.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-70 years.
2. Diagnosis of Alcoholic hepatitis based on NIAAA criteria
3. MELD 20-35
4. Willing to follow up

Exclusion Criteria:

1. Patients with hepatic/ extra hepatic malignancies
2. Patients with contraindications to steroids
3. Patients who are critically ill and are admitted to the ICU
4. Patient who have severe extra hepatic organ failure
5. Patients who are HBsAg +, HIV+
6. If female of childbearing potential: known pregnancy, or unwilling to practice anticontraceptive measures
7. Patients who are on current treatment with prednisone and/or immunosuppressive me.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of MMF versus steroid therapy in improving short-term (28 day) survival outcomes in patients with alcoholic hepatitis | 28 days

SECONDARY OUTCOMES:
MDF Score in alcoholic hepatitis in both the groups at 28 days and 90 days. | 28 days and 90 days.
Number of patients with adverse events in both the groups. | 28 days and 90 days.
To compare the efficacy of MMF versus steroid therapy in improving long-term (90 day) survival outcomes in patients with alcoholic hepatitis | 28 days and 90 days.
To see molecular biomarkers like Interleukin (IL 6), Interleukin(IL 1) and their response to both the therapies. | 28 days and 90 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided